CLINICAL TRIAL: NCT02836353
Title: The Metabolic Consequences of Gastrointestinal Surgery
Brief Title: Metabolic Consequences of Gastrointestinal Surgery
Acronym: MaS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reached scientific goals, further recruitment would not further advance the findings of study.
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Geoffrey Roberts, Clinical Research Associate, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A093993
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Gastrectomy; Oesophagectomy; Dumping Syndrome; Hypoglycaemia
MeSH Terms: conditions — Dumping Syndrome; Hypoglycemia | interventions — Somatostatin; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Observational only (No Intervention): Oral glucose tolerance test, neurocognitive questionnaire tasks only.
- Somatostatin (Experimental): Oral glucose tolerance test after 100mcg Somatostatin
  Interventions: Drug: Somatostatin
- Antibiotics (Experimental): Oral glucose tolerance test after treatment of small intestinal bacterial overgrowth
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Somatostatin — Single dose of short acting Somatostatin (100mcg) pre Oral glucose tolerance test
  Arms: Somatostatin
Drug: Rifaximin — 1 week course of 400mg three times daily (TDS) pre Oral glucose tolerance test
  Arms: Antibiotics

SUMMARY:
Surgery on the gastrointestinal (GI) tract results in profound changes to the metabolic profile. This is well described, including the rapid resolution of diabetes seen after bariatric surgery. The underlying pathophysiology, and incidence in lean patients undergoing surgery for cancer, is somewhat less described. The investigators plan to assess the symptomatic and glycaemic profile, as well as causative pathways, for metabolic symptoms in patients after surgery on the GI tract. The investigators will use glucose tolerance tests, physiological challenges with somatostatin analogues and antibiotics, and assess tissue transcriptomic changes.

DETAILED DESCRIPTION:
The role of the gut hormone axis in glucose control is of significant interest due to its proven translational impact in diabetes management. It is also significantly altered by gastric surgery, a procedure that can lead to deleterious symptoms (dumping syndrome) in lean, non-diabetic patients. The investigators will study a unique cohort of young, lean patients undergoing surgery for the prevention of gastric cancer, as well as patients undergoing surgery for gastric and oesophageal cancer, to further understand the regulation and pathophysiological role of the gut hormone axis. The prophylactic patient population will be recruited from the pool of patients with a genetic mutation conferring a high lifetime risk of gastric cancer (Hereditary Diffuse Gastric Cancer) for whom Addenbrooke's Hospital provides a national clinical service. The investigators aim to define the causative physiological pathways for dumping syndrome in this group and expand our body of knowledge of gut hormones and their role in glucose homeostasis and eating behaviour.

It has been suspected for some years that surgery has more profound physiological effects than simple anatomical rearrangement, however recent developments in bariatric surgery have brought this to the fore. The era of surgical treatment of peptic ulcer disease resulted in a large cohort of patients undergoing gastric surgery and suffering post-operative dumping symptoms. These include symptoms attributed to hypovolaemia immediately after a meal, followed by hypoglycaemia within a few hours. There was a significant hiatus in the study of dumping syndrome after the decline of surgery for ulcer disease in the 1980s. The major improvement in long-term survival after surgery for oesophageal and gastric cancer seen in the 21st Century, coupled with the identification of high risk familial cohorts who now undergo prophylactic gastrectomy, has led to a growing cohort of long-term survivors after gastrectomy. This presents the significant challenge of defining and managing the ongoing, quality of life-limiting metabolic consequences of gastrointestinal surgery. The late dumping symptoms suffered by this patient cohort include paradoxical post-prandial hypoglycaemia, likely resulting from an excessive insulin response to particular components of ingested food.

There is also a population of patients undergoing oesophagectomy for malignant or pre-malignant conditions of the oesophagus, who receive post-operative nutrition through a feeding tube sited through the abdominal wall and entering the jejunum approximately 1 metre from its origin. This group of patients suffer similar metabolic changes to those undergoing gastrectomy, and provide a unique opportunity to study the differential response to nutrients administered orally or more distally. This could elucidate the role of any proximal gut hormones in glucose homeostasis.

The recent expansion in understanding of the metabolic effects of surgery has largely been driven by the study of bariatric (better termed metabolic) surgery. It is well known that Roux-en-Y gastric bypass (RYGB) can result in early remission of diabetes in 85% of cases and elevated levels of gut hormones such as glucagon-like peptide 1 (GLP-1), but there is considerable debate around whether the gut hormones changes contribute to the reductions in plasma glucose and appetite after surgery. Whereas studies in rodent models appear to indicate that gut hormones are largely redundant after bypass surgery, data from humans strongly support the idea that increased post-prandial GLP-1 and Peptide YY (PYY) levels underlie improvements in insulin secretion and reduced appetite. Studies from bariatric cohorts are confounded by the requirement for dietary restriction before surgery and massive weight loss after surgery.

Multiple studies have measured the baseline and stimulated levels of circulating gut hormones after RYGB in obese subjects. Elevated levels of GLP-1 and PYY and reduced levels of ghrelin have been reported in most studies, and variable results have been found for glucose-dependent insulinotropic peptide (GIP), cholecystokinin (CCK) and pancreatic polypeptide (PP).

Fewer studies have addressed the changes in gut hormone secretion after gastrectomy in lean subjects. Limited studies have demonstrated changes in GLP-1 secretion. Literature on the experimental approach to dumping pathways is largely limited to case reports or small series but indicates a role for the glucose-insulin axis.

The role of gut microbiota in determining host metabolism is a topical area of interest, following discoveries that lean and obese phenotypes can be transferred by gut microbial transplantation in rodent models. Despite the excitement surrounding this area, it remains a highly controversial research field, and the extent to which the human microbiome influences energy metabolism is hotly debated. A variety of microbial metabolites, including short chain fatty acids and indole, however, modulate gut hormone secretion, and likely contribute to basal gut hormone release in the fasting state. An interesting question that has not previously been addressed is whether gut hormone secretion becomes more dependent on microbial metabolism after bypass surgery, either because resident colonic bacteria are supplied with an increased load of fermentable nutrients, or because of increased bacterial growth in the proximal intestine (small intestinal bacterial overgrowth). It is, however, well established that microbial metabolism is altered in some post-surgical patients, as assessed non-invasively by the appearance of raised hydrogen or methane levels in exhaled breath. It is also possible that the differing pool of bacteria between people may contribute to a varied metabolic phenotype - it is therefore important to characterise the microbiome to assess changes arising due to surgery or antibiotic treatment.

Beyond the purely physiological effects of surgery, there is an increasing understanding that removal of the stomach or oesophagus has a profound effect on a person's appetite and eating behaviour. This likely results from the central action of gut derived hormones, and is an area of significant interest in the obesity field. Anecdotally, post-gastrectomy patients frequently report minimal appetite and significant changes in their food preferences. At present, this has not been characterised in a scientifically rigorous fashion. A variety of tools exist to assess the motivation and impulsivity of a person's relationship to food in a non-invasive fashion, which can be administered from home, or as an adjunct to a gut hormone secretion test.

Previous studies from the investigators' group and beyond have demonstrated that L cells, the prime enteroendocrince cells (EECs) secreting GLP-1, directly sense glucose uptake and have receptors for bile acids and short chain free fatty acids (bacterial fermentation products of carbohydrates). Each of these pathways could theoretically contribute to the enteroendocrine detection of ingested carbohydrate, but the relative importance of the different sensory mechanisms before, as well as after, GI surgery is unknown.

Overall, this proposed study of gut hormone secretion and metabolism in the lean population will define the causative pathways of dumping syndrome and provide a model for the study of post-operative gut hormone changes without the confounding effects of massive weight loss. In turn, this will expand knowledge of the physiological pathways underlying gut hormone secretion and their role in glucose homeostasis, with the potential to offer new therapeutic and research targets in diabetes and obesity care, as well as in this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone previous oesophageal or gastric resection

Exclusion Criteria:

* Age <18
* Recent history of untreated anaemia
* Donated blood in preceding 16 weeks
* Lack capacity to read and retain information about study
* Have a known allergy to interventional agent
* Have received a course of antibiotics in preceding two months
* Be on medication that interacts with intervention
* Have a history of C. difficile colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Severity of hypoglycaemia during glucose tolerance test as measured by plasma glucose levels | Glucose tolerance test immediately after drug intervention

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey P Roberts, MA BM BCh, Principal Investigator — University of Cambridge; Fiona M Gribble, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts GP, Kay RG, Howard J, Hardwick RH, Reimann F, Gribble FM. Gastrectomy with Roux-en-Y reconstruction as a lean model of bariatric surgery. Surg Obes Relat Dis. 2018 May;14(5):562-568. doi: 10.1016/j.soard.2018.01.039. Epub 2018 Feb 3. PMID 29548882
- [Result] Roberts GP, Larraufie P, Richards P, Kay RG, Galvin SG, Miedzybrodzka EL, Leiter A, Li HJ, Glass LL, Ma MKL, Lam B, Yeo GSH, Scharfmann R, Chiarugi D, Hardwick RH, Reimann F, Gribble FM. Comparison of Human and Murine Enteroendocrine Cells by Transcriptomic and Peptidomic Profiling. Diabetes. 2019 May;68(5):1062-1072. doi: 10.2337/db18-0883. Epub 2019 Feb 7. PMID 30733330
- [Result] Larraufie P, Roberts GP, McGavigan AK, Kay RG, Li J, Leiter A, Melvin A, Biggs EK, Ravn P, Davy K, Hornigold DC, Yeo GSH, Hardwick RH, Reimann F, Gribble FM. Important Role of the GLP-1 Axis for Glucose Homeostasis after Bariatric Surgery. Cell Rep. 2019 Feb 5;26(6):1399-1408.e6. doi: 10.1016/j.celrep.2019.01.047. PMID 30726726